CLINICAL TRIAL: NCT01647737
Title: A Natural Formulation for Patients Diagnosed With Xerostomia
Brief Title: Green Tea Lozenges for the Management of Dry Mouth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Scott DeRossi, Chairman, Diagnostic Sciences, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHSU Lozenge Xerostomia Study
Record Dates: First submitted 2012-05-14; First posted 2012-07-24 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Xerostomia; Sjogren Syndrome; Dry Mouth
Keywords: Xerostomia; Sjogren syndrome; dry mouth
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome | interventions — Xylitol; Aspartame

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MighTeaFlow (Active Comparator): 4-6 times daily lozenge containing green tea, jaborandi extracts, and 500 mg xylitol for 8 weeks
  Interventions: Dietary Supplement: MighTeaFlow
- Xylitol (Active Comparator): 4-6 times daily lozenge containing jaborandi extract, and 500 mg xylitol for 8 weeks
  Interventions: Dietary Supplement: Xylitol

INTERVENTIONS:
Dietary Supplement: MighTeaFlow — 4-6 times daily
  Other Names: Green Tea Lozenge
  Arms: MighTeaFlow
Dietary Supplement: Xylitol — 4-6 times daily
  Other Names: Aspartame
  Arms: Xylitol

SUMMARY:
The goal of this proposal is to investigate the effectiveness of a Medical College of Georgia patent pending formulation of natural plant extracts on patients with xerostomia. The major component of this formulation is green tea extract with a defined composition of polyphenols. Epidemiological studies suggest that phytochemicals in green tea possess beneficial effects on autoimmune and inflammatory diseases. Thus far, there is little evidence to indicate any marked and direct immunomodulatory effect of green tea on T or B lymphocytes. However, there is considerable evidence for green tea polyphenols (GTPs), major phytochemicals found in green tea extract, having properties consistent with effects on cells of tissues that would be protective towards local inflammation.

DETAILED DESCRIPTION:
Patients with subjective complaints of xerostomia will be given a screening questionnaire to complete. If they meet the criteria on this screening form, the research coordinator will be notified and will meet with the patient either immediately or at a scheduled follow-up appointment. The research coordinator will review the information and then explain the details of the study to the patient and obtain informed consent. Once the patient has signed the informed consent, the research coordinator will collect the demographic, medical history, and contact information from the patient. Any information missing will be noted for follow-up investigation by the research coordinator. If a subject is of child bearing age, they will be asked to complete a urine pregnancy test prior to enrollment.[a] First appointment -Screening, consent. [b]Follow appointments- review, then Patients will do VAS questionnaire, QOL questionnaire, Sialometry will be done measuring unstimulated whole saliva and Stimulated whole saliva for 5 min each.

ELIGIBILITY:
Inclusion Criteria:

1. A complaint of dry mouth as assessed by a response of 30mm or greater on a Dry Mouth Visual Analog Scale (VAS)
2. Clinical Diagnosis of primary or secondary Sjogren's syndrome.
3. Over the age of 18.
4. Taking less than three drugs associated with causing xerostomia or salivary gland hypofunction.
5. Willing to use natural novel topical dry mouth products.
6. Prior minor salivary gland biopsy and serology from Sjogren's Syndrome/Xerostomia work-up.
7. Willing to return for all study-associated visits.
8. Able to read, understand, and sign the informed consent.

Exclusion Criteria:

1. Have received radiation to the head and neck region.
2. Unable to read and understand the consent form.
3. On greater than three drugs associated with xerostomia or salivary gland hypofunction.
4. Require dento-alveolar surgery or extensive dental treatment during the course of the study.
5. Require hospitalization for any medical problem during the course of the study.
6. Unable to take green tea leaf extract and/or pilocarpus jaborandi leaf extract and/or xylitol because of allergy
7. Uncontrolled medical conditions that require changes in medication during the course of the study.
8. Regularly consume green tea and/or components of pilocarpus jaborandi.
9. Are pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott S De Rossi, DMD, Principal Investigator — GHSU
Locations (1):
- GHSU Center for Oral Medicine, Augusta, Georgia, United States

REFERENCES:
- [Derived] De Rossi SS, Thoppay J, Dickinson DP, Looney S, Stuart M, Ogbureke KU, Hsu S. A phase II clinical trial of a natural formulation containing tea catechins for xerostomia. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Oct;118(4):447-454.e3. doi: 10.1016/j.oooo.2014.06.015. Epub 2014 Jul 5. PMID 25240992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential candidates were identified from a pool of previously diagnosed subjects and new subjects referred to the Clinical Center for Oral Medicine, School of Dentistry, Georgia Regents University
Pre-assignment Details: Subjects had a diagnosis of Xerostomia
Groups:
- Green Tea Lozenge: GTP
  Green tea lozenge: 4-6 times daily
- Placebo: Xylitol lozenge 4 - 6 times daily
Period: Overall Study
Arm/Group | Green Tea Lozenge | Placebo
Started | 30 | 30
Completed | 26 | 25
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Population: Consented subjects diagnosed with Xerostomia and meeting all inclusion exclusion criteria
Groups:
- Placebo: Xylitol
  Green tea lozenge: 4-6 times daily
- Total: Total of all reporting groups
Arm/Group | Green Tea Lozenge | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 13 | 14 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Salivary Flow From Baseline
Description: Change in salivary flow in Xerostomic patients using Green tea lozenges
Time Frame: 8 weeks
Population: Enrolled subjects completing 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Green Tea Lozenge | Placebo
Number analyzed (Participants) | 26 | 27
ml/min
  Week 0 | 0.17 (0.051) | 0.10 (0.278)
  Week 8 | 0.66 (0.168) | 0.04 (0.142)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 27 months
Arm/Group | MighTeaFlow | Xylitol
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MighTeaFlow (N=30) | Xylitol (N=30)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — itching and scratchiness in the throat

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No